CLINICAL TRIAL: NCT02281916
Title: Safety Study of P28GST Treatment in Crohn's Disease Patients, a Multicenter Phase 2 Clinical Trial
Brief Title: Safety Study of P28GST Treatment in Crohn's Disease Patients
Acronym: ACROHNEM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: National Research Agency, France (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013_02; 2013-000595-15 (EudraCT Number)
Record Dates: First submitted 2014-10-28; First posted 2014-11-04 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2018-06

CONDITIONS: Crohn's Ileocolitis
Keywords: Crohn disease; Immunotherapy; Helminth antigen
MeSH Terms: conditions — Crohn Disease | interventions — Immunotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- P28GST treatment (Experimental): P28GST as a parasite enzyme
  Interventions: Drug: P28GST

INTERVENTIONS:
Drug: P28GST — 3 injections of 100 µg of P28GST within 3 months (one injection per month)
  Other Names: immunotherapy

SUMMARY:
This multicenter phase 2 clinical trial is designed to assess safety of P28GST (protein 28 Kd glutathion S Transferrase), aiming to control inflammation in moderate Crohn's Disease (CD), before or after intestinal resection surgery. P28GST is a parasite enzyme molecule from Schistosoma with potent immunogenic and anti-oxidant properties. Based on experimental evidence of its anti-inflammatory properties, the investigators hypothesized that administration of P28GST could protect against recurrence after intestinal resection surgery in CD.

DETAILED DESCRIPTION:
To carry out this study, 24 moderate CD patients will be enrolled in a safety phase 2a study. CD patients will be included after intestinal resection surgery or in moderate Crohn's Disease (CD). Drug therapy will consisted in 3 injections of 100 µg of P28GST within 3 months (one injection per month). The main objective of this study is to follow-up monthly rate and seriousness of adverse events during one year. Secondary objectives are to control immunologic and inflammatory blood and tissue markers, appearance or not of a clinical recurrence assessed by CDAI (Crohn Disease Activity Index).

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of ≥18 years at inclusion.
* Subjects with ileal or ileo-colic CD without fistula
* Subjects operated or not
* CDAI score < 220
* no concomitant treatment excepted salicylates
* Women of child bearing potential must be negative for pregnancy prior to study enrolment
* contraceptive means : females of childbearing potential as well as males are required to use adequate contraceptive methods for 6 months starting at the inclusion, i;e 4 months after the 3rd injection .
* No tobacco consumption (end date of tobacco consumption 8 days before surgery).
* Signed consent form
* French social security coverage.

Exclusion Criteria:

* Subject who use of azathioprine, anti-TNF (Tumor Necrosis Factor), methotrexate, Vedolizumab, Ustekinumab and other immunosuppressors for 8 weeks before first injection of P28GST
* Subject who use of corticosteroids for 15 days before first injection of P28GST
* Subject with history of vaccine hyper sensitivity or allergy.
* Subject with any other clinical manifestation determined by the investigator
* Subject wih AIDS, B or C hepatitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2014-03; Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Number of participants wtih adverse events as a measure of safety and tolerability | up to one year
  Clinical and blood markers change from baseline

SECONDARY OUTCOMES:
Main immunologic and inflammatory blood and tissue markers. | up to one year
Appearance or not of a clinical recurrence assessed by CDAI (Crohn Disease Activity Index) and confirmed by a morphologic examination. | up to one year
Intestinal microbiota | at inclusion, at 4 month , at 12 month
  Evolution of bacterial species by genomic analysis

CONTACTS AND LOCATIONS:
Overall Officials: Dominique DEPLANQUE, MD, PhD, Study Chair — Lille University Hospital
Locations (5):
- France (5):
  - Centre hospitalier, Amiens
  - Centre Hospitalier de Boulogne, Boulogne-sur-Mer
  - Centre Hospitalier Dunkerque, Dunkirk
  - CHRU, Hôpital Claude Huriez, Lille
  - Centre Hospitalier,, Valenciennes

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Foligne B, Ple C, Titecat M, Dendooven A, Pagny A, Daniel C, Singer E, Pottier M, Bertin B, Neut C, Deplanque D, Dubuquoy L, Desreumaux P, Capron M, Standaert A. Contribution of the Gut Microbiota in P28GST-Mediated Anti-Inflammatory Effects: Experimental and Clinical Insights. Cells. 2019 Jun 12;8(6):577. doi: 10.3390/cells8060577. PMID 31212833